CLINICAL TRIAL: NCT04594889
Title: Comparison of Sirolimus vs Paclitaxel Drug Eluting Balloon for Below-the-knee Angioplasty in Critical Limb Ischemia
Acronym: DebateBTKDuell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Francesco Liistro, Cardiovascular Intervention Director, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N° 1916-22/09/2020
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Critical Limb Ischemia; Drug Effect
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus (Experimental): Sirolimus eluting balloon will be inflated in the target vessel after optimal balloon angioplasty for at least 2 minutes
  Interventions: Procedure: angioplasty
- Paclitaxel (Active Comparator): Paclkitaxel eluting balloon will be inflated in the target vessel after optimal balloon angioplasty for at least 2 minutes
  Interventions: Procedure: angioplasty

INTERVENTIONS:
Procedure: angioplasty — Balloon releasing a drug inflated in the target vessel
  Other Names: PTA

SUMMARY:
The objective of this study is to compare the remote patency of paclitaxel versus sirolimus eluting balloons in patients with CLI undergoing tibial artery revascularization. Patients will be randomized 1:1 to Paclitaxel eluting balloon (Litos, ACOTEC ltd) or sirolimus eluting balloon (Magic touch, Concept Medical) after optimal balloon angioplasty. The primary endpoint of the study is the late luminal loss at 6 months angiography. Secondary endpoint are major amputation, clinically driven target lesion revascularization and vessel reocclusion (duplex) at 12 months.

DETAILED DESCRIPTION:
Critical ischemia of the limb is considered one of the most severe clinical scenario of atherosclerotic disease involving the lower limb because it is associated with a high degree of mortality and morbidity. Below the knee arterial disease is the basis of critical limb ischemia (CLI). It is generally characterized by the involvement of multiple tibial arteries, long lesions and high rate of hronic total occlusions. Percutaneous treatment of tibial arteriopathy is characterized by high restenosis (70%). The advent of the drug-eluting strategy has led to a reduction in the restenosis of the femoral and tibial district with paclitaxel eluting devices. Data are not yet available on sirolimus eluting devices, both for the femoropopliteal and tibial districts. The objective of this study is to compare the remote patency of paclitaxel (Lithos) vs. the sirolimus (magic touch) eluting balloons in patients with CLI undergoing tibial artery revascularization.

The study will enroll only patients with optimal balloon angioplasty defined by angiographic and ultrasound criteria in order to avoid biases related to potentially unbalanced suboptimal angioplasty results in both groups. The patients will be followed by either interventionalists as well as diabetic foot specialists in order to optimize their surveillance for lesion healings and vessel patency and reduced dropout.

Participating

Centers Cardiovascular disease department (San Donato Hospital, Arezzo, Italy) O.U. Cardiology (San Iacopo Hospital, Pistoia, Italy) O.U. Cardiology (San Giuseppe Hospital, Empoli, Italy) O.U Hemodynamics (A.O.U.C. Careggi, FlorenCe, Italy)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years
2. CLI Rutherford class 4-6.
3. Stenosis or occlusion with length >= 4 cm involving a tibial artery
4. Presence of angiographic distal runoff to the foot (stage 1-2a-2b of the Kawarada classification)
5. Presence of optimal angioplasty result defined as residual stenosis < 50%, absence of flow limiting dissection, absence of vessel perforation, absence of distal embolization by angiography and biphasic or triphasic flow at ultrasoud evaluation of the target vessel

Exclusion Criteria:

1. Known allergy to one of the drugs in the study
2. Contraindications to antiplatelet therapy
3. Life expectancy less than 1 year
4. Major amputation planned before angiography
5. Inability to obtain informed consent -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-10-14 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Late Luminal Loss (LLL) | 6 months
  LLL will be measured in the treated segment obtained subtracting the minimal lumen diameter at 6-month angiographic follow.up with minimal lumen diameter post intervention

SECONDARY OUTCOMES:
Major limb amputation | 12 months
  amputation of target limb that requires a prostesis for standing and walking
Clinically driven target lesion revascularization | 12 months
  repeat intervention of the target segment due to vessel restenosis documented by angiography and the presence of symptoms as follows:
  1. non healing ulcer
  2. rest pain of the treated limb
Target vessel occlusion (TVO) | 12 months
  TVO will be documented by duplex ultrasond examination

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Liistro, MD, Principal Investigator — Ospedale San Donato
Locations (1):
- Ospedale San Donato, Arezzo, AR, Italy

IPD SHARING:
Plan to Share IPD: No